CLINICAL TRIAL: NCT05635578
Title: The Effect of Reiki Applicatıon on Sleep and Qualıty of Life in Epılepsy Patıents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/30-34
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Sleep; Life Quality
MeSH Terms: interventions — Sleep; Quality of Life

STUDY DESIGN:
Intervention Model Description: reiki
Who Masked: Participant
Masking Description: Single (Participant) sleep, life quality
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (Experimental): reiki will be aplicated
  Interventions: Behavioral: sleep
- Control (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Behavioral: sleep — reiki
  Other Names: life quality
  Arms: Experimental:

SUMMARY:
After the general period of positive social adjustments, epilepsy is in a high life cycle to control seizures. During seizures in epilepsy, patients' quality of life and antiepileptic life span can be seen in daily life such as daily life and daily awakenings.

Reiki, which has been proven by studies in health problems such as fatigue and pain; an energy that can be unblocked or applied in a non-applicable way can benefit from a therapy that can be applied by touch or remotely, without negative effects. In the literature, reiki applied to epilepsy patients has sleep and quality of life. This thesis is planned to do research on sleep and living areas of reiki applied to epilepsy patients.

DETAILED DESCRIPTION:
This research; It will be carried out on a voluntary basis with the treatment of 60 patients with epilepsy, 30 of which will be tested, 30 of which will be comprehensive, from the University of Fır Hospital Neurology Clinic Polyclinic and those over 18 years of age, who can communicate adequately, who have psychiatric problems, who are in the last six body mind, who can control the phone, who will come to the scale, who will come to sleep. The study will be a pretest-posttest controlled group study. Data; Patient Information Form will be collected with Pittsburgh Sleep Quality Scale, Quality of Life in Epilepsy Scale. The control method will not interfere. If we try, first the application places and the way of doing it will be shown. Administration through 4 weeks, first consecutive week; 1 session face-to-face 30-45 minutes, then 3 sessions of 21 minutes of training, 2 sessions of 21 minutes of training in the other 3 training courses, a total of 4 weeks 10. For face-to-face reiki; A room will be used inside the hospital. Reiki to 7 different chakras to be taken in the first session. For the other sessions, before the application, all will be called and informed about the reiki will be sent, and then he will apply reiki from a distance for 21 minutes by using the training and reiki symbols. The scales will be reapplied by the researcher, either face to face or face to face, during the experiment and 4 weekends to be controlled. Finally, there will be a significant difference between the pretest and the son test.

ELIGIBILITY:
* be over 18 years old
* Ability to communicate adequately
* Absence of psychiatric problems
* Not having received body-mind therapy (yoga, reiki, massage, meditation) in the last six months
* Volunteering to participate in the research
* Own a phone
* Having a scale score of greater than 5 according to the Pittsburgh Sleep Quality Scale
* Not using sleeping pills 4.4.2. Exclusion Criteria from Research
* being under the age of 18
* Having trouble communicating
* Having a psychiatric problem
* Having received body-mind therapy (yoga, reiki, massage, meditation) in the last six months
* Not being willing to participate in the research
* Not having a phone
* Having a scale score of less than and/or equal to 5 on the Pittsburgh Sleep Quality Scale
* Using sleeping pills

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 1 hours later
  The Pitssburgh sleep quality index, developed by Buysse et al. in 1989, is used to evaluate the quality of sleep, the amount of sleep, the presence and severity of sleep disorders in the last month. Agargun et al. They adapted PUKI to Turkish in 1996.There are seven components in the scale. These; subjective sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), use of sleeping pills (component 6) and daytime dysfunction (component 3) 7) stop. The evaluation score of each item is between 0-3, and the total score obtained at the end of the evaluation is between 0-21. A total score of 5 and less than 5 defines good sleep, and a total score of more than 5 defines poor sleep
Quality of Life Scale in Epilepsy | 1 hours later
  The Quality of Life Scale for Patients with Epilepsy was developed by Vickrey et al. in 1993. Mollaoğlu et al. carried out the validity and reliability studies of this scale in Turkey in 2015. The scale includes 7 sub-dimensions. These sub-dimensions are; anxiety about seizures (5 items), effects of drugs (3 items), energy/fatigue (4 items), emotional well-being (5 items), cognitive function (6 items), social function (5 items), total quality of life (2 items) ) and an additional item that evaluates the total health status, a total of 31 items. Scale scoring is in the range of 0-100. High score indicates higher quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Gülcan B Turan, Elâzığ, Merkez, Turkey (Türkiye)